CLINICAL TRIAL: NCT01032655
Title: The Efficacy of Susceptibility Test -Driven Sequential Therapy as the Third Line Therapy for Refractory Helicobacter Pylori Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Attending physician, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200901042M
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; sequential therapy; susceptibility-driven; rescue; levofloxacin; clarithromycin; salvage; treatment failure; those who fail from two standard eradication therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sequential, susceptibility guided (Experimental): single arm
  Interventions: Drug: susceptibility test guided sequential therapy

INTERVENTIONS:
Drug: susceptibility test guided sequential therapy — susceptibility test driven sequential therapy D1- D7 Nexium ,40mg, bid Amolin, 1gm bid D8-14 Nexium ,, 40mg, bid Flagyl, 500mg, bid
  plus either one of the following
  1. Klaricid, 500 mg, bid
  2. Cravit, 250 mg, bid
  3. Tetracycline, 500 mg, bid

SUMMARY:
Background: Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection could reduce the occurence or recurrence of these diseases. However, it was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy. About 15-30% of patient would fail from second line therapy and need to be rescued with third line therapy. The commonly used salvage regimens include (1) Bismuth based quadruple therapy (combined with ranitidine or PPI plus two antibiotics) (2) Levofloxacin or moxifloxacin or rifabutin based triple therapy. However, Bismuth is not available in many countries and the administration method is complex. Its usage is limited by the high pill number and low compliance rate. In recent years, the concept of sequential therapy has been advocated in the treatment of H. pylori infection. The regimen includes a PPI plus amoxicillin for five days, followed by a PPI plus clarithromycin and metronidazole for another five days. The eradication rate in the first line treatment of sequential therapy had been reported to be as high as 90%. More importantly, it has been demonstrated that the eradication rate among patients with clarithromycin-resistant strains could be as high as 89%. According to the Maastricht III consensus meeting, it was recommended that susceptibility test should be done for patients who failed two treatments. Therefore, we aimed to assess the efficacy of susceptibility test driven sequential therapy as the third line therapy for those who fail from two standard eradication therapies.

Methods: This will be a multi-center, open labeled pilot study

1. Patients:

   * Open labeled, non-comparative pilot study
2. Testing for H. pylori infection:

   * Before salvage treatment:

   either (1) any two positive of CLO test, histology, and culture or (2) a positive C13-UBT will be considered as failure of previous eradication treatment EGD with gastric biopsy will be done for H. pylori culture and susceptibility test
   * After salvage treatment: C13-UBT will be used to assess the existence of H. pylori after 2nd or 3rd line salvage therapy
3. Treatment regimens and assignment:

   * D1-7: Nexium (40 mg, bid), Amolin (1 gm, bid)
   * D8-14: Nexium (40 mg, bid), Flagyl (500 mg, bid) plus either one of the following according to antibiotic susceptibility test (1) Klaricid, 500 mg, bid or (2) Cravit, 250 mg, bid or (3) Tetracycline, 500 mg, bid
4. Outcome Measurement:

   * Primary End Point: Eradication rate will be evaluated according to Intent-to-treat (ITT) and per-protocol (PP) analyses
   * Secondary End Point: the eradication rate according to antibiotic susceptibility before salvage therapy

ELIGIBILITY:
Inclusion Criteria:

1. aged greater than 20 years who have persistent H. pylori infection after two treatments and are willing to receive third line rescue regimens.

Exclusion Criteria:

1. children and teenagers aged less than 20 years,
2. history of gastrectomy,
3. gastric malignancy, including adenocarcinoma and lymphoma,
4. previous allergic reaction to antibiotics (Amolin, Klaricid, Cravit) and prompt pump inhibitors (esomeprazole),
5. contraindication to treatment drugs,
6. pregnant or lactating women,
7. severe concurrent disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Eradication rate will be evaluated according to Intent-to-treat (ITT) and per-protocol (PP) analyses | 2009/04/20

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Ming Liou, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Liou JM, Chen CC, Chang CY, Chen MJ, Fang YJ, Lee JY, Chen CC, Hsu SJ, Hsu YC, Tseng CH, Tseng PH, Chang L, Chang WH, Wang HP, Shun CT, Wu JY, Lee YC, Lin JT, Wu MS; Taiwan Helicobacter Consortium. Efficacy of genotypic resistance-guided sequential therapy in the third-line treatment of refractory Helicobacter pylori infection: a multicentre clinical trial. J Antimicrob Chemother. 2013 Feb;68(2):450-6. doi: 10.1093/jac/dks407. Epub 2012 Oct 25. PMID 23099849